CLINICAL TRIAL: NCT01629992
Title: Preoperative Counseling in Cholecystectomy. A Randomized Trial
Brief Title: Preoperative Counseling in Cholecystectomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of Mato Grosso (Other)
Responsible Party: Principal Investigator, Jose Eduardo de Aguilar-Nascimento, Chairman Professor, Federal University of Mato Grosso
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: preopcounseling; 697/CEP-HUJM/09 (Other: HUJM Research Ethics Committee)
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Vomiting; Nausea; Postoperative Pain; Feeling
Keywords: Vomiting; Nausea; Postoperative pain; Feeling
MeSH Terms: conditions — Vomiting; Nausea; Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preoperative counseling (Experimental): The intervention group received preoperative counseling by both orally and written. A written leaflet containing information was provided to each patient of this group.
  Interventions: Other: Preoperative counseling
- Control (No Intervention): The control group received no preoperative counseling either oral or written.

INTERVENTIONS:
Other: Preoperative counseling — The intervention group received preoperative counseling by both orally and written. A written leaflet containing information was provided to each patient of this group.
  Other Names: Preoperative information
  Arms: Preoperative counseling

SUMMARY:
The investigators examined whether a written plus verbal preoperative counseling for patients undergoing open cholecystectomy would improve perioperative symptoms such as nausea, vomiting and pain.

DETAILED DESCRIPTION:
This was a randomized, single-blinded, clinical study carried out at the Julio Muller University Hospital (Mato Grosso State, Brazil). This study was conducted according to the guidelines laid down in the Declaration of Helsinki and all procedures involving human subjects/patients were approved by the hospital Research Ethics Committee registered under number 697/CEP-HUJM/09. Written informed consent was obtained from all patients.

Except for the preoperative counseling which was received only by the intervention group, all patients received the same protocol of perioperative care.

The main endpoint of the study was the presence and the intensity of postoperative symptoms such as nausea, vomiting and pain. A questionnaire containing a visual analogue scale (VAS) was applied 24h after the operation to measure the intensity of postoperative pain, nausea and the well-being. The VAS consisted of a horizontal line, 100 mm in length, anchored by word descriptors at each end to represent the lowest and the highest intensity of all the symptoms analyzed. The patient was asked to mark in the straight line the point that most likely represents the symptom at the moment. The VAS score of each individual was determined by measuring in millimeters from the left end of the line to the point marked. The questions were: "how severe was your pain during this period of 24h after the operation?", "how severe was the intensity of your nausea during this period of 24h after the operation? ", and "how great is your well-being at the present moment". For the first two questions the words at each end of the line were "no pain" and "severe pain", and "no nausea" and "severe nausea". For the well-being question the words were "no well-being" and "greatest well-being". The Vomiting was also recorded as a categorical variable (yes or no). The length of stay and postoperative complications were also collected.

ELIGIBILITY:
Inclusion Criteria:

* adult age (18-65 years-old),
* both sexes and
* candidates for an elective open cholecystectomy

Exclusion Criteria:

* having diabetes mellitus,
* chronic kidney failure,
* chronic liver disease,
* serum bilirubin > 2 mg/dL,
* body mass index (BMI) > 35 kg/m2,
* American Anesthesiologists Association (ASA) score > 3,
* gastro-esophageal reflux,
* gastroparesis or intestinal obstruction.

Patients with any non-compliance with the study protocol, who had the choledochus opened or associated operations, who experienced severe intraoperative complications (any type of shock, cardiac arrest or coagulations problems) or experienced prolonged (> 4 h) operative time were also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2009-01; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 24h after operation
  A questionnaire containing a visual analogue scale (VAS) was applied 24h after the operation to measure the intensity of postoperative pain, nausea and the well-being. The VAS consisted of a horizontal line, 100 mm in length, anchored by word descriptors at each end to represent the lowest and the highest intensity of all the symptoms analyzed. The patient was asked to mark in the straight line the point that most likely represents the symptom at the moment. The VAS score of each individual was determined by measuring in millimeters from the left end of the line to the point marked.

SECONDARY OUTCOMES:
Episodes of vomiting | During the first 24h after surgery
  Number of episodes of vomiting occurring until 24h after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Jose Aguilar-Nascimento, MD, PhD, Principal Investigator — Federal University of Mato Grosso
Locations (1):
- Hospital Universitario Julio Mullar, Cuiabá, Mato Grosso, Brazil